CLINICAL TRIAL: NCT05848440
Title: A Phase I Randomised Single-blind Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD9550 Following Single Ascending Dose Administration to Healthy Participants
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD9550 Following Single Ascending Dose Administration to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D8460C00001; 2022-003308-34 (EudraCT Number)
Record Dates: First submitted 2023-03-31; First posted 2023-05-08 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: Non-alcoholic steatohepatitis (NASH); Liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Intervention Model Description: Placebo-control
Who Masked: Participant, Investigator
Masking Description: The participant and the Clinical Unit staff will remain blinded during the dosing phase of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental): Participants will be administered single ascending SC doses of AZD9550 or a placebo.
  Interventions: Drug: AZD9550; Drug: Placebo
- Part B (Experimental): Participants will be administered one SC dose of AZD9550 or a placebo.
  Interventions: Drug: AZD9550; Drug: Placebo
- Part C (Experimental): Participants will be administered one IV dose of AZD9550 or a placebo.
  Interventions: Drug: AZD9550; Drug: Placebo

INTERVENTIONS:
Drug: AZD9550 — Participants will be administered AZD9550 subcutaneously.
  Arms: Part A; Part B
Drug: AZD9550 — Participants will be administered AZD9550 intravenously.
  Arms: Part C
Drug: Placebo — Participants will be administered matching volumes of placebo subcutaneously or intravenously.

SUMMARY:
This is a Phase I Randomised Single-blind Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD9550 Following Single Ascending Dose Administration to Healthy Participants.

DETAILED DESCRIPTION:
This study will be a Phase I, First-In-Human (FIH), randomised, single-blind, placebo-controlled, single ascending dose (SAD), sequential group study in healthy male and female participants of non- childbearing potential performed at a single study centre.

The study consists of 3 parts:

* Part A: SAD (up to 5 dose levels) of AZD9550 administered subcutaneous (SC) in healthy participants.
* Part B: 1 dose level of AZD9550 administered SC in healthy participants of Japanese descent.
* Part C: 1 dose level of AZD9550 administered intravenous (IV) in healthy participants.

The study will comprise of:

* A Screening Period of maximum 28 days.
* A Treatment Period during which participants will be resident at the Clinical Unit from 2 days before (Day -2) investigational medicinal product (IMP]) administration (Day 1) until at least 7 days (168 hours; Day 8) after IMP administration.
* Weekly out-clinic visits on Days 15, 22, 29, and 36.
* A Follow-up Visit 6 weeks (Day 43) after the IMP dose.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* Healthy male and female participants aged 18 to 55 years.
* Females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit, must not be lactating, and must be of non childbearing potential, confirmed at the Screening Visit by fulfilling one of the following criteria:

  1. Postmenopausal defined as amenorrhoea for at least 12 months or more following cessation of all exogenous hormonal treatments and Follicle stimulating hormone (FSH) levels in the postmenopausal range.
  2. Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* Have a Body mass index (BMI) between 18 and 30 kg/m^2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive at Screening and admission.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of Investigational medicinal product (IMP).
* Any laboratory values with the following deviations at Screening and admission:

  1. Alanine aminotransferase > Upper limit of normal (ULN)
  2. Aspartate aminotransferase > ULN
  3. eGFR < 60 mL/min/1.73m2 (to be calculated using CKD-EPI formula)
  4. White blood cell count < LLN
  5. Hemoglobin < LLN
  6. Neutrophil Count <1.5 × 10*9/L
* Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results other than those described under exclusion criterion number 4, as judged by the Investigator.
* Any positive result at Screening for serum hepatitis B surface antigen, hepatitis C antibody and Human immunodeficiency virus (HIV).
* Abnormal vital signs, after 10 minutes supine rest at Screening.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting Electrocardiogram (ECG) and any clinically important abnormalities in the 12 lead ECG that may interfere with the interpretation of QTc interval changes, including abnormal ST T wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9550.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest.

Note: participants consented and screened, but not randomised in this study or a previous Phase I study, are not excluded.

* Judgment by the Investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the Screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
* Participants with a medical history of Medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome (MEN 2), or a baseline serum calcitonin at or above 50 ng/L.
* Any condition that would have interfered with the evaluation of the IMP or interpretation of participant safety or study results.
* Participants who are unable to consume in full the MMTT (Mixed meal tolerance test - Ensure Plus 200 mL).
* Participants with a medical history of MTC (Medullary thyroid carcinoma) or MEN 2 (multiple endocrine neoplasia syndrome), or a baseline serum calcitonin at or above 50 ng/L.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) | Throughout the study (up to 6 months)
  The safety and tolerability of AZD9550 following SC administration of single ascending doses to healthy participants, SC administration of a single dose to Japanese participants, and IV administration of a single dose to healthy participants will be assessed.

SECONDARY OUTCOMES:
Area under concentration time curve from time 0 to infinity (AUCinf) | Day 1 until Day 43 (follow-up visit)
  The AUCinf of AZD9550 following SC administration of single ascending doses to healthy participants, SC administration of a single dose to Japanese participants, and IV administration of a single dose to healthy participants will be assessed.
Area under concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | Day 1 until Day 43 (follow-up visit)
  The AUClast of AZD9550 following SC administration of single ascending doses to healthy participants, SC administration of a single dose to Japanese participants, and IV administration of a single dose to healthy participants will be assessed.
Maximum observed concentration (Cmax) | Day 1 until Day 43 (follow-up visit)
  The Cmax of AZD9550 following SC administration of single ascending doses to healthy participants, SC administration of a single dose to Japanese participants, and IV administration of a single dose to healthy participants will be assessed.
Incidence of Anti-Drug Antibodies (ADAs) | Day 1 until Day 43 (follow-up visit)
  The immunogenicity of AZD9550 following SC and/or IV administration of AZD9550 will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/